CLINICAL TRIAL: NCT03692845
Title: Minimally Invasive Versus Open Transforaminal Lumbar Interbody Fusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Hatem Ahmed Mohammed, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6272829
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Spinal Fusion
Keywords: spine fusion; minimally invasive surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- O-TLIF group (Other): Spinal fusion ,Transforaminal lumbar interbody fusion procedure will be performed through open surgery.
  Interventions: Procedure: Transforaminal Lumbar Interbody Fusion either open or minimally invasive
- MI-TLIF group (Other): Spinal fusion,Transforaminal lumbar interbody fusion procedure will be performed through minimally invasive surgery using a tubular retractor.
  Interventions: Procedure: Transforaminal Lumbar Interbody Fusion either open or minimally invasive

INTERVENTIONS:
Procedure: Transforaminal Lumbar Interbody Fusion either open or minimally invasive — Spinal fusion procedure through the intervertebral foramen

SUMMARY:
A study that compares between Open TLIF and Minimally invasive TLIF regarding patients' functional status(Oswestry Disability index)as a primary outcome measure.

DETAILED DESCRIPTION:
The first randomized controlled trial comparing minimally invasive TLIF and open TLIF.

ELIGIBILITY:
Inclusion Criteria:

* Adults more than 18 years of age and less than 65 years of age..
* Degenerative or isthmic spondylolithesis Grade 1,2 and 3.
* Recurrent Symptomatic recurrent lumbar disc prolapsed with or without evident neural compression.
* Single level pathology involving L2-3, L3-4, L4-5 and or L5-S1.
* Symptoms not responding to conservative treatment for at least 3 months.

Exclusion Criteria:

* Previous spinal fusion or instrumentation.
* Spinal tumours, infection and fractures.
* Patients with severe osteoporosis
* BMI more than 35.
* Non-ambulant patients and patients with severe preoperative neurological affection (Cauda Equina Syndrome)
* Patients not willing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability index(Arabic version) 1 month | 1 month
  an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain.

SECONDARY OUTCOMES:
• Fusion rate as assessed by Bridwell fusion score. | 1 year
  Grade I is defined as fusion with remodelling and trabeculae present; Grade II is an intact graft with incomplete remodelling and no lucency present; Grade III is an intact graft with potential lucency at the cranial or caudal end; Grade IV is absent fusion with collapse/resorption of the graft.

IPD SHARING:
Plan to Share IPD: No